CLINICAL TRIAL: NCT04083560
Title: A Comparison of Two Different Doses of Maternal B12 Supplementation in Improving Infant B12 Deficiency and Neurodevelopment
Acronym: MATCOBIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sitaram Bhartia Institute of Science and Research (Other)
Collaborators: Public Health Foundation of India (Other); Paropakar Matenity and Women's Hospital, Kathmandu, Nepal (Unknown); University College, London (Other)
Responsible Party: Principal Investigator, Dr Jitender Nagpal, Senior Consultant and Head of the Department, Sitaram Bhartia Institute of Science and Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MATCOBIND 2018
Record Dates: First submitted 2019-09-02; First posted 2019-09-10 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Vitamin B 12 Deficiency
MeSH Terms: conditions — Vitamin B 12 Deficiency | interventions — Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Group A Intervention: 360 pregnant women will receive 250 mcg of B-12 daily orally from 1st trimester to 6 months postpartum
  Interventions: Drug: Vit B12
- Control group (Active Comparator): Group B- Control: 360 pregnant women will receive 50 mcg of B-12 daily orally from 1st trimester to 6 months post partum
  Interventions: Drug: Vit B12

INTERVENTIONS:
Drug: Vit B12 — Vitamin B12 250mcg

SUMMARY:
Supplementation with Iron and folate have been part of a worldwide strategy targeting anaemia and neural tube defects for many years. However, vitamin B12 deficiency has received much less attention. High prevalence of deficiency in mothers in the antenatal period and in their infants, has been documented. Multiple case series document the neurological consequences of severe deficiency and their reversal with B-12. Trials on the subject are limited and those available have either used an ineffective dose or for a short duration.

Therefore, we propose this randomised controlled trial to compare the efficacy of two different doses (pharmacological and preventive) of maternal Vitamin B-12 supplementation in improving infant B12 deficiency and neurodevelopment. We propose to undertake a multi-centric trial in India and Nepal given the high prevalence of deficiency reported from these countries and to allow a wider socio-demographic spectrum (Pay-for-service hospital catering to middle income populace from India and a free-care public hospital catering to lower income groups from Nepal). We will recruit 720 vegetarian, pregnant women from the antenatal clinics of the Indian and Nepalese centres at their first antenatal visit. Elderly primi mothers, taking B12 supplementation, multiple gestations, chronic medical conditions, anticipating moving out of the city, treated for infertility or with known psychological illnesses will be excluded. In Stage 1, recruited mothers will be randomized into 2 equal groups (360 each). Group 1-Daily 250 μg Vitamin B12 supplementation. Group 2-Daily 50 μg Vitamin B12 supplementation. B-12 will be started in 1st trimester and continue up to 6 months post-partum. In Stage 2, the birth and post-delivery course of the new-born will be monitored and documented for any morbidity. At 9 months, the neurodevelopmental, complementary feeding and home environment will be assessed and infant B12 status will be determined.

The two groups will be compared for the primary (neurodevelopment) and secondary outcomes (biochemical parameters in mother and infant). The results of this study will be used to generate scientific evidence on whether B-12 should be supplemented in vegetarian pregnant women with a view to preventing B-12 deficiency and its neurodevelopmental consequences in the infant.

ELIGIBILITY:
Inclusion Criteria:

* <12 weeks gestation

Vegetarian mothers

Exclusion Criteria:

1. Mothers already on B12 supplementation
2. Women with multiple gestation, those diagnosed with chronic medical conditions (diabetes mellitus, hypertension, heart disease, neurological disease or thyroid disease), and those who tested positive for hepatitis B, HIV or syphilis (associated with prematurity, IUGR and other neonatal morbidities which could influence neurodevelopment)
3. Women who anticipate moving out of the city before/ after delivery
4. Women treated for infertility
5. Women with known psychological illnesses including depression

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 708 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
Infant neurodevelopment | 9 Month of infant age
  Developmental Assessment Scale for Indian Infant (modified Bayleys scale) measured as average of motor and mental scores

SECONDARY OUTCOMES:
Biochemical B12 status of mother | At recruitment
  Change in B12 status of mother between first and third trimester
Biochemical B12 status of infant | 9 months of infant age
  Biochemical B12 status of infant at nine months postpartum

OTHER OUTCOMES:
Mean Haemoglobin of infants | 9 months of infant age
  Haemoglobin of infants in grams per deciliter
Infant weight | 9 months of infant age
  Infant weight in kilograms
Infant length | 9 months of infant age
  Infant Length in cms
Infant head circumference | 9 months of infant age
  Infant Head circumference in cms

CONTACTS AND LOCATIONS:
Locations (2):
- Sitaram Bhartia Institute of Science and Research, New Delhi, National Capital Territory of Delhi, India
- Rajendra Pant, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nagpal J, Mathur MR, Rawat S, Nagrath D, Lee C, Singhal A, Heys M, Cortina Borja M, Augustin K, Gautam J, Pant R, Swabey L, Lakhanpaul M. Efficacy of maternal B12 supplementation in vegetarian women for improving infant neurodevelopment: protocol for the MATCOBIND multicentre, double-blind, randomised controlled trial. BMJ Open. 2020 May 25;10(5):e034987. doi: 10.1136/bmjopen-2019-034987. PMID 32457078